CLINICAL TRIAL: NCT00402272
Title: SPIRIT V: A Clinical Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System in the Treatment of Patients With de Novo Coronary Artery Lesions
Brief Title: SPIRIT V: Post-marketing Evaluation of the XIENCE V® Everolimus Eluting Coronary Stent System in Europe
Acronym: SPIRIT V
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Ellen Travis, Abbott Vascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-369
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; stents; Angioplasty; coronary artery disease; total coronary occlusion; coronary artery restenosis; stent thrombosis; vascular disease; myocardial ischemia; coronary artery stenosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): XIENCE V® Everolimus Eluting Coronary Stent System
  Interventions: Device: XIENCE V® Everolimus Eluting Coronary Stent

INTERVENTIONS:
Device: XIENCE V® Everolimus Eluting Coronary Stent — Drug eluting stent implantation stent in the treatment of coronary artery disease.
  Other Names: XIENCE V® Everolimus Eluting Coronary Stent System

SUMMARY:
The purpose of this Clinical Evaluation is a continuation in the assessment of the performance of the XIENCE V® Everolimus Eluting Coronary Stent System (XIENCE V® EECSS) in the treatment of patients with de novo coronary artery lesions.

DETAILED DESCRIPTION:
The SPIRIT V Clinical Evaluation consists of two concurrent studies,the Diabetic Sub-Study and the Registry.

The SPIRIT V Registry is a prospective, single arm, multi-center registry evaluating performance of the XIENCE V® EECSS in real-world use, per its Instruction For Use (IFU). 2,700 patients will be enrolled in the SPIRIT V Registry.

The long term safety and efficacy of the XIENCE V EECSS have been demonstrated in the SPIRIT FIRST trial up to 5 years, the SPIRIT II trial up to 4 years, and in the SPIRIT III Randomized Control Trial (RCT) up to 3 years. In addition, these pre-approval studies have shown low rates of Target Vessel Failure and Major Adverse Cardiac Events (MACE) that were observed to plateau or gradually decline after about 1 year and were consistently lower than the comparator arm of each study. This benefit in MACE is sustained for up to 5 years and is also independent of the first year results.

The post approval SPIRIT V study demonstrated that the use of the XIENCE EECSS in complex lesions in a real-world population resulted in 1 year MACE, Stent Thrombosis and Target Lesion Revascularization rates that are comparable to those of the previously mentioned pre-approval studies which included patients with more restricted inclusion / exclusion criteria.

Therefore, based on existing data from these trials, Abbott Vascular has decided to discontinue further follow up in the SPIRIT V Registry study after 2 years.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the XIENCE V® EECSS and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure, as approved by the appropriate Medical Ethics Committee of the respective clinical site
* evidence of myocardial ischemia
* acceptable candidate for coronary artery bypass graft (CABG) surgery
* undergo all CIP-required follow-up examinations
* artery morphology and disease is suitable to be optimally treated with a maximum of 4 planned XIENCE V® EESCC
* target lesions must be de novo lesions
* target vessel reference diameter must be between 2.5 mm and 4.0 mm by visual estimate
* target lesion ≤ 28 mm in length by visual estimate

Exclusion Criteria:

Patient is already participating in another device or drug study or has completed the follow-up phase of another study within the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2700 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
SPIRIT V Registry: Adjudicated Composite rate of All Death, Myocardial Infarction (MI) and Target Vessel Revascularization (TVR) . | at 30 days

SECONDARY OUTCOMES:
SPIRIT V Registry: Acute Success (Clinical Procedure Success) | Acute
SPIRIT V Registry: Adjudicated Stent Thrombosis (Confirmed/definite, Probable, Possible) | at 30 days, 1 and 2 years
SPIRIT V Registry: Adjudicated Revascularizations (TLR/TVR/any Revascularization) | at 30 days, 1 and 2 years
SPIRIT V Registry: Adjudicated Composite rate of Cardiac Death, MI attributed to the target vessel and TLR | at 30 days, 1 and 2 years
SPIRIT V Registry: Adjudicated Composite rate of All Death, any MI and TVR | at 30 days, 1 and 2 years
SPIRIT V Registry: Adjudicated Composite rate of All Death, any MI and any Revascularization(TLR/TVR/non TVR) | at 30 days, 1 and 2 years
SPIRIT V Registry: Acute Success (Clinical Device Success) | Acute

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Grube, MD, Principal Investigator — The Heart Center, Siegburg, Germany; Upendra Kaul, MD, Principal Investigator — Fortis Hospital, New Delhi, India
Locations (93):
- Salzburger Landeskliniken, Salzburg, Austria
- Belgium (5):
  - UCL St Luc, Brussels
  - ULB Erasmus Hospital, Brussels
  - UZ Gent, Ghent
  - Hopital St Joseph, Gilly
  - Clinique St. Luc - Bouge, Namur
- Canada (7):
  - Foothills Medical Center, Calgary
  - CHUM Hotel Dieu Hospital, Montreal
  - Montreal Heart Institute, Montreal
  - University of Ottawa Heart Institute, Ottawa
  - Hôpital Laval, Québec
  - Sunnybrook and Women's College, Toronto
  - University health Network - Toronto Gen Hospital, Toronto
- China (5):
  - Fuwai Hospital, Beijing
  - Prince of Wales Hospital, Hong Kong
  - PYNEH, Hong Kong
  - Queen Elizabeth, Hong Kong
  - Zhongshan Hospital, Shanghai
- Univerzity Hospital Hradec Králové, Karlove, Czechia
- France (7):
  - C.H.U. - Hopital Michallon, Grenoble
  - CHU Lille - Hôpital Cardiologique, Lille
  - NCN - Nouvelle Cliniques Nantaises, Nantes
  - Hopital privé Les Fransiscaines, Nîmes
  - La pitié Salpétrière, Paris
  - Polyclinique St Laurent, Rennes
  - C.C.N., Saint-Denis
- Germany (7):
  - Kerckhoff Klinik GmbH, Bad Nauheim
  - Herzzentrum, Bernau
  - Universitätsklinikum, Heidelberg
  - Lukas Krankenhaus Neuss, Neuss
  - Herzzentrum Siegburg GmbH, Siegburg
  - Universitätsklinikum Ulm, Ulm
  - Helios Klinikum Wuppertal, Wuppertal
- Onassis Cardiac Center, Athens, Greece
- India (8):
  - Krishna Heart Institute, Ahmedabad
  - Apollo Hospital, Chennai
  - Institute of Cardiovascular Disease M.M.M., Chennai
  - All India Institute of Medical Science - AIIMS, Delhi
  - Fortis Hospital, Delhi
  - B M Birla, Kolkata
  - Kailash Hospital, New Delhi
  - Ruby Hall Clinic, Pune
- Ireland (2):
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (3):
  - Hadassah-Hebrew University Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Ichilov Medical Center, Tel Aviv
- Italy (11):
  - Azienda USL 8, Arezzo
  - Azienda Ospedaliera Riuniti, Bergamo
  - Emodinamica Azienda Spedali Civili, Brescia
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - Emodinamica Cardiologia Azienda ULSS 12 Veneziana, Ospedale Civile Umberto 1, Mestre
  - Ospedale Civile, Mirano
  - Azienda Ospedaliera di Padova, Padua
  - IRCCS Policlinico San Matteo, Pavia
  - Ospedale San Filippo Neri, Roma
  - Policlinico A. Gemelli, Roma
  - Azienda Ospedaliera S. Gdi Dio Salerno, Salerno
- Malaysia (2):
  - Institute Jantung Negara, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Netherlands (3):
  - Medisch Centrum Alkmaar, Alkmaar
  - Catharina ZH Eindhoven, Eindhoven
  - Maasstad Ziekenhuis, Rotterdam
- Christchurch Hospital, Christchurch, New Zealand
- Portugal (3):
  - Hospital Garcia da Orta, Lisbon
  - Hospital Santa Cruz, Lisbon
  - Hospital Santa Marta, Lisbon
- National University Hospital, Singapore, Singapore
- South Africa (2):
  - Sunninghill Hospital, Johannesburg
  - Vergelegen Clinic, Vergelegen
- Spain (14):
  - Hospital del Mar, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Universitari de Bellvigte, Barcelona
  - Trias Y Pujol, Barcelona
  - Valle Hebron, Barcelona
  - Puerta del Mar, Cadiz
  - Policlinica Gipuzkoa, Donostia / San Sebastian
  - Clinico San Carlos, Madrid
  - Hospital Puerta de Hierro, Madrid
  - La Paz, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Son Dureta, Palma de Mallorca
  - Marques de Valdecilla, Santander
  - Meixoeiro-Medtec, Vigo
- Uppsala Univ. Hospital, Uppsala, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Thailand (2):
  - Bhumibol Adulyadej Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
- United Kingdom (5):
  - Wessex Cardiac Unit, Southampton, Southampton
  - Royal Sussex County, Brighton, Brighton
  - Glenfield Hospital, Leicester
  - King's College Hospital, London
  - Wythenshawe Hospital, Manchester

REFERENCES:
- [Derived] Genereux P, Rutledge DR, Palmerini T, Caixeta A, Kedhi E, Hermiller JB, Wang J, Krucoff MW, Jones-McMeans J, Sudhir K, Simonton CA, Serruys PW, Stone GW. Stent Thrombosis and Dual Antiplatelet Therapy Interruption With Everolimus-Eluting Stents: Insights From the Xience V Coronary Stent System Trials. Circ Cardiovasc Interv. 2015 May;8(5):e001362. doi: 10.1161/CIRCINTERVENTIONS.114.001362. PMID 25940520
- [Derived] Ringel RE, Gauvreau K, Moses H, Jenkins KJ. Coarctation of the Aorta Stent Trial (COAST): study design and rationale. Am Heart J. 2012 Jul;164(1):7-13. doi: 10.1016/j.ahj.2012.04.008. Epub 2012 Jun 20. PMID 22795276
- [Derived] Grube E, Chevalier B, Guagliumi G, Smits PC, Stuteville M, Dorange C, Papeleu P, Kaul U, Dzavik V. The SPIRIT V diabetic study: a randomized clinical evaluation of the XIENCE V everolimus-eluting stent vs the TAXUS Liberte paclitaxel-eluting stent in diabetic patients with de novo coronary artery lesions. Am Heart J. 2012 May;163(5):867-875.e1. doi: 10.1016/j.ahj.2012.02.006. Epub 2012 Apr 11. PMID 22607866